CLINICAL TRIAL: NCT04373525
Title: Substance Misuse To Psychiatric Disorders for Cannabis-Prospective Evaluation on Cognitive Function and Its Associated Genetic Vulnerability in Cannabis Users (SToP-C-PeCoG)
Brief Title: Prospective Evaluation on Cognitive Function and Its Associated Genetic Vulnerability in Cannabis Users
Acronym: SToP-C_PeCoG
Status: Enrolling by invitation | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Albert Kar-Kin Chung, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 20-189
Record Dates: First submitted 2020-04-23; First posted 2020-05-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Cannabis Use; Neurocognitive Dysfunction; Genetic Predisposition
Keywords: Cannabis; Cognition; Genetics
MeSH Terms: conditions — Cognition Disorders; Genetic Predisposition to Disease; Marijuana Abuse | interventions — Genome-Wide Association Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Genome analysis — Venous blood will be obtained for later genome analysis

SUMMARY:
Most of the studies assessing Cannabis Use Disorder (CUD) and neurocognitive functions are cross-sectional without examining the longitudinal changes in neurocognitive function at a within-subject level with respect to the continuum of cannabis use behavior, or mainly studying on the acute cannabis effect. As for the Genome-wide Association studies, the population analyzed for addressing the underlying genetic susceptibility between neurocognitive functions and/or cannabis use or CUD were almost exclusively based on African- or European- American samples or other Caucasian subjects, and thus generalizability to Chinese or to the non-Caucasian population definitely demands more studies.

With the upsweeping statistical figures of cannabis use in Hong Kong and Asia, and the substantial falls in the perceived risk and personal disapproval from using cannabis amongst young abusers, coinciding the global advocacy of de-criminalizing cannabis and the increased availability of recreational cannabis worldwide, it is reasonable to predict that there will be a further upsurge in numbers of all aged cannabis users in Hong Kong as in the other part of the world. Therefore, the SToP-C-PeCoG study proposed here as a prospective study in assessing the longer term changes in neurocognitive functions and the associated genetic risks for those repeated and active cannabis users without psychiatric co-morbidity is definitely warranted. The PeCoG study will not only provide the scientific evidence to further unveil the harmful effects on neurocognitive functions for those self-perceived "healthy" users, but also help to raise the public awareness and to improve the understandings to the long-term detrimental effects of cannabis amongst users and non-users. Furthermore, it will provide a chance to study the associated genetic risks for cannabis abusers, in particular in the Asian minority and Chinese, on CUD and poorer neurocognitive outcomes, with genetic vulnerability being generalizable to the local population in Asia.

The current study hypothesises that cannabis abusers have neurocognitive function decline over time, and genetic vulnerability is associated with cannabis abusers who have poorer neurocognitive outcomes or with the severity of CUD.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 - 60 years old at the time of enrolment
* Able to read and communicate in English and/or Chinese
* Able to give informed consent
* Using cannabis or marijuana as the primary psychoactive substance of abuse
* Repeated and Active cannabis users as defined by Structured Clinical Interview for DSM-5 Disorders

Exclusion Criteria:

* Age <16 years old
* Unable to read English or Chinese
* Unable to give informed consent
* Had been diagnosed with other Substance Related Disorders, except for Tobacco Use Disorders due to the known frequent comorbid use for cannabis users (12)
* Currently taking regular prescribed psychiatric medications, including antipsychotics, antidepressants, mood stabilizers, anti-epileptics, benzodiazepines, hypnotics, and anti-cholinergic medications.
* Had been diagnosed with DSM-5 disorders, other than Cannabis Use and related disorders

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 16-60 years old cannabis users
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 18 months
  Subject assessed with a maximum score of 30. Those who score 26 or below will consider to have mild cognitive impairment
Frontal Assessment Battery | 18 months
  Subject who scores 12 or below will be considered having frontal dysexcutive function
Wechsler Memory Scale | 18 months
  Subject will be assessed with the scale for their immediate, delayed, visual and auditory memory
Genome analysis | Each subject only need to have venous blood test once 1 day within their 18-months study period
  venous blood test will be done on consented subject for genome analysis for associated single nucleotide polymorphisms on 4 related chromosomes identified from literature associated with cannabis use disorder and neurocognitive impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
data without identifiable